CLINICAL TRIAL: NCT07019792
Title: Effect of Different Rotary Files Systems on Post-operative Pain and Bacterial Reduction in Lower Single Canal Posterior Teeth With Necrotic Pulp: Prospective Double Blinded Clinical Trial
Brief Title: Postoperative Pain and Bacterial Reduction in Oval Canals After Instrumentation With Different Noval Rotary Files Systems
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ruba Mustafa, Professor associate, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20230408; 20230408 (Other Grant/Funding Number: Jordan University of Science and Technology)
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Bacterial Count Reduction in Oval Canal After Rotary Instrumentation With Different Systems; Post-operative Pain After Rotary Instrumentation of Oval Canal With Different Systems
Keywords: post operative pain; Protaper Ultimate; Hyflex EDM; XP rsie; TruNatomy; Bacterial; Oval canal
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Multifile system: Protaper Ultimate (Experimental)
  Interventions: Other: Protaper ultimate
- Multiple files systems:TruNatomy (Experimental)
  Interventions: Other: Truanatomy file system
- Single file system: Hyflex EDM (Experimental)
  Interventions: Other: Hyflex EDM
- Single file system: Xp shaper rise (Experimental)
  Interventions: Other: Xp shaper rise

INTERVENTIONS:
Other: Protaper ultimate — Using Protaper Ultimate file system for canal preperation
  Arms: Multifile system: Protaper Ultimate
Other: Truanatomy file system — Using Truanatomy file system for canal preperation
  Arms: Multiple files systems:TruNatomy
Other: Hyflex EDM — Using Hyflex file system for canal preperation
  Arms: Single file system: Hyflex EDM
Other: Xp shaper rise — Using XPshaper rise system for canal preperation
  Arms: Single file system: Xp shaper rise

SUMMARY:
Postoperative pain after endodontic treatment can affect a patient's quality of life. It is reported that debris extrusion after the instrumentation technique can influence postoperative pain. As a result, the aim of this clinical trial is to compare the recent rotary systems (TruNatomy, ProTaper Ultimate, Hyflex EDM and XP- rise rotary files systems) in terms of apical extrusion defined by post-operative pain and their role in reducing the bacterial count inside the canal

DETAILED DESCRIPTION:
One hundred and twenty lower premolar teeth will be included in the study(n=120). Teeth will be randomly assigned to one of the 4 groups(n=30). Preoprative pain will be recorded before root canal treatment. Postoperative pain will be recorded using visual analogue scale (VAS) at 6 hours,12 hours, 1day, 2 days, 3 days, 4 dayse and five days after the root canal treatment. Bacterial count before and after instrumentation will be determined using culturing methods to determine the bacterial count reduction.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit
* Age ranges from 18-65 year
* Restorable teeth
* Necrotic teeth and symptoms free
* Lower premolars teeth (single canal posterior teeth)
* Necrotic pulps

Exclusion Criteria:

* Medically compromised
* Non-restorable teeth
* Open apex canal
* The past 12-hour history of analgesic intake before treatment.
* Patients with a history of antibiotics intake in the last 3 months before treatment.
* Pregnant females.
* Symptomatic patient.
* Pulpal diagnosis is not necrotic pulp.
* Retreatment cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | at 6hours,12 hours, 24 hours, 2 days, 3 days, 4 days and five days after the root canal treatment
  Postoperative pain will be recorded using Visual Analogue Scale (VAS) at 6hours,12 hours, 24 hours, 2 days, 3 days, 4 days and five days after the root canal treatment Visual Analogue Scale (VAS) ranges from 0-10, the lower number the better outcome.
  0= no pain 1-3= mild pain 4-6= moderate pain 7-10= sever pain
Bacterial count reduction | Sample will be collected before and directly after canal prepeartion
  Bacterial count sample will be collected before and after canal prepeartion

CONTACTS AND LOCATIONS:
Locations (1):
- Ruba Mustafa, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No